CLINICAL TRIAL: NCT01403402
Title: Congenital Muscle Disease Patient and Proxy Reported Outcome Study
Brief Title: Congenital Muscle Disease Study of Patient and Family Reported Medical Information
Acronym: CMDPROS
Status: Recruiting | Type: Observational
Sponsor: Cure CMD (Other)
Responsible Party: Sponsor
Other Study IDs: CMDPROS1
Record Dates: First submitted 2011-07-26; First posted 2011-07-27 (Estimated); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Congenital Muscular Dystrophy With ITGA7 (Integrin Alpha-7) Deficiency; Alpha-Dystroglycanopathy (Congenital Muscular Dystrophy and Abnormal Glycosylation of Dystroglycan With Severe Epilepsy); Alpha-Dystroglycanopathy (Congenital Muscular Dystrophy With Fatty Liver and Infantile-onset Cataract Caused by TRAPPC11 Mutations); Alpha-Dystroglycanopathy (Congenital Muscular Dystrophy With Hypoglycosylation of Dystroglycan); Alpha-Dystroglycanopathy (Congenital Muscular Dystrophy With Hypoglycosylation of Dystroglycan and Epilepsy); Alpha-Dystroglycanopathy (Dystroglycanopathy, Congenital With or Without Mental Retardation (Formerly MDC1C)); Alpha-Dystroglycanopathy (Fukuyama CMD); Alpha-Dystroglycanopathy (LGMDR09 FKRP Related (Formerly LGMD2I)); Alpha-Dystroglycanopathy (LGMDR11 POMT1 Related (Formerly LGMD2K)); Alpha-Dystroglycanopathy (LGMDR13 FKTN Related (Formerly LGMD2M)); Alpha-Dystroglycanopathy (LGMDR14 POMT2 Related (Formerly LGMD2N)); Alpha-Dystroglycanopathy (LGMDR15 POMGnT1 Related (Formerly LGMD2O)); Alpha-Dystroglycanopathy (LGMDR19 GMPPB Related (Formerly LGMD2T)); Alpha-Dystroglycanopathy (LGMDR20 ISPD Related (Formerly LGMD2U)); Alpha-Dystroglycanopathy (LGMDR24 POMGnT2 Related); Alpha-Dystroglycanopathy (Muscle Eye Brain Disease (MEB)); Alpha-Dystroglycanopathy (Walker Warburg Syndrome (WWS)); Choline Kinase B Receptor - CHKB; Collagen VI Related Disorders; Collagen XII Related Disorders; Congenital Muscular Dystrophy Not Otherwise Specified (Including Merosin Positive); Congenital Muscular Dystrophy With Cataracts and Intellectual Disability (MDCCAID); Congenital Muscular Dystrophy With Joint Hyperlaxity; Congenital Muscular Dystrophy With Rigid Spine Related to ACTA1; Emery-Dreifuss Muscular Dystrophy; GOLGA2-related Congenital Muscle Dystrophy With Brain Involvement; LMNA Related Disorders; Merosin Deficient CMD (Full or Partial); Nesprin Related MD (SYNE1); SELENON Related Disorders (Previously Known as SEPN1); SELENON Related Myopathy (Aka SEPN1); Telethonin CMD; Congenital Myasthenic Syndrome; Limb-Girdle Muscular Dystrophy; LGMDD01 - DNAJB6 (Formerly LGMD1D); LGMDD05 - Collagen VI Related Bethlem Myopathy (Dominant); LGMDR07 - Telethonin (TCAP) Related (Formerly LGMD2G); LGMDR08 - TRIM Related (Formerly LGMD2H); LGMDR09 - FKRP Related (Formerly LGMD2I); LGMDR10 - Titin (TTN) Related (Formerly LGMD2J); LGMDR11 - POMT1 Related (Formerly LGMD2K); LGMDR13 - Fukutin (FKTN) Related (Formerly LGMD2M); LGMDR14 - POMT2 Related (Formerly LGMD2N); LGMDR15 - POMGnT1 Related (Formerly LGMD2O); LGMDR16 - DAG1 Related Dystroglycanopathy (Formerly LGMD2P); LGMDR17 - Plectin (PLEC) Related (Formerly LGMD2Q); LGMDR18 - TRAPPC11 Related (Formerly LGMD2S); LGMDR19 - GMPPB Related (Formerly LGMD2T); LGMDR20 - ISPD Related (Formerly LGMD2U); LGMDR22 - Collagen VI Related Bethlem Myopathy (Recessive); LGMDR23 - LAMA2 Related; LGMDR24 - POMGnT2 Related
Keywords: Congenital Muscular Dystrophy; Congenital Myopathy; Neuromuscular Diseases; Musculoskeletal Diseases
MeSH Terms: conditions — Muscular Dystrophy, Congenital, Due To Integrin Alpha-7 Deficiency; Epilepsy; Walker-Warburg Syndrome; Wieacker syndrome; Intellectual Disability; Muscular Dystrophy, Emery-Dreifuss; Myasthenic Syndromes, Congenital; Muscular Dystrophies, Limb-Girdle; Muscular Dystrophy, Limb-Girdle, Type 2G; Muscular Dystrophy, Limb-Girdle, Type 2M; Myotonia Congenita; Neuromuscular Diseases; Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Congenital Muscle Disease: The congenital muscle diseases include congenital muscular dystrophy, congenital myopathy, congenital myasthenic syndrome and bridge into the limb girdle/late onset spectrum. For data collection and analysis, subtype specific reports will be generated. True incidence of the congenital muscle diseases is unknown.

SUMMARY:
The Congenital Muscle Disease Patient and Proxy Reported Outcome Study (CMDPROS) is a longitudinal 10 year study to identify and trend care parameters, adverse events in the congenital muscle diseases using the Congenital Muscle Disease International Registry (CMDIR) to acquire necessary data for adverse event calculations (intake survey and medical records curation). To support this study and become a participant, we ask that you register in the CMDIR. You can do this by visiting www.cmdir.org. There is no travel required.

The registry includes affected individuals with congenital muscular dystrophy, congenital myopathy, and congenital myasthenic syndrome and registers through the late onset spectrum for these disease groups. The CMDIR was created to identify the global congenital muscle disease population for the purpose of raising awareness, standards of care, clinical trials and in the future a treatment or cure. Simply put, we will not be successful in finding a treatment or cure unless we know who the affected individuals are, what the diagnosis is and how the disease is affecting the individual.

Registering in the CMDIR means that you will enter demographic information and complete an intake survey. We would then ask that you provide records regarding the diagnosis and treatment of CMD, including genetic testing, muscle biopsy, pulmonary function testing, sleep studies, clinic visit notes, and hospital discharge summaries.

Study hypothesis:

1. To use patient and proxy reported survey answers and medical reports to build a longitudinal care and outcomes database across the congenital muscle diseases.
2. To generate congenital muscle disease subtype specific adverse event rates and correlate with key care parameters.

DETAILED DESCRIPTION:
The Congenital Muscle Disease Patient and Proxy Reported Outcome Study (CMDPROS) is a longitudinal 10 year observational study to identify care and trend key care parameters and adverse events in the congenital muscle diseases using the Congenital Muscle Disease International Registry (CMDIR). The CMDIR registers individuals with and without genetic confirmation who have been given a clinical diagnosis of congenital muscular dystrophy, congenital myopathy, and congenital myasthenic syndrome, or myofibrillar myopathy, through the limb girdle/late onset spectrum.

Identifying care parameters and adverse events in the rare genetic neuromuscular diseases can be difficult. Care is fragmented, genetic confirmation may not be prioritized by the medical community or covered by medical insurance and patients are scattered globally with potential challenges aggregating data across centers. Natural history studies are currently being launched. However, potential biases to participation include recruitment of the less severely affected patients given difficulty traveling secondary to a medically fragile condition. There is currently no treatment for these conditions; though optimizing and standardizing care and care delivery can promote significant gains in quality of life and survival. Identifying disease specific care parameters and correlating those parameters with adverse event rates will not only contribute to the development of evidence based guidelines but inform clinically meaningful outcomes for future clinical trials.

Study hypothesis:

1. To use patient and proxy reported survey answers and medical reports to build a longitudinal care and outcomes database across the congenital muscle diseases.
2. To generate congenital muscle disease subtype specific adverse event rates and correlate with key care parameters.

Primary outcome is survival measured from date of birth to date of death. Primary outcome will be analyzed by congenital muscle disease subtype and maximal ambulatory status achieved.

Secondary outcomes include disease specific adverse event rates including rates of hospitalization, rates of antibiotic use, rates of pulmonary infections, pneumothorax, atelectasis, aspiration and adverse complaints including bloating, constipation, chest pain, dyspnea assessed by a validated breathing assessment, vomiting and nausea and difficulty eating. Patient and proxy hospitalization, pneumothorax and atelectasis reports will be confirmed by obtaining hospital discharge summaries. Additional secondary outcomes include ejection fraction (relevance subtype specific), forced vital capacity in liters, weight, Rapid Eye Movement (REM) sleep apnea hypopnea index and mean oxygen saturation during REM and total sleep study, age, gender, type of treatment center location (national referral center, tertiary care hospital, community hospital), gastrostomy tube, total number of fractures and Tscore/Zscore of hip and spine on DEXA scans.

Preliminary studies may focus on specific congenital muscle disease subtypes and use retrospective data collection through registry, survey monkey and telephone interviews to assess adverse event rates over last month and last year to limit recall bias. Prospective enrollment of same study participants over 12 months will assess monthly rates of adverse events and complaints. A preliminary study, CMD PROADE (Patient and Proxy Reported ADverse Event Rates) is planned in 2 congenital muscular dystrophy subtypes: Collagen 6 Myopathy and LAMA 2 Related CMD.

De-identified data from CMDIR will be made available for IRB approved natural history studies in the congenital muscle diseases.

ELIGIBILITY:
Inclusion Criteria:

Alpha 7/Alpha 9 Integrin Related Myopathy Collagen VI Related Myopathy (Ullrich through Bethlem CMD) Alpha-Dystroglycan Related Muscular Dystrophy (Dystroglycanopathy, WWS, MEB, Fukuyama, FKRP, LGMD2I, LGMD2K, LGMD2M, LGMD2N, LGMD2O) Choline Kinase B Receptor Emery-Dreifuss Muscular Dystrophy (EDMD, LGMD1B, LMNA, Emerin, FHL1, SYNE1, SYNE2, TMEM43) LAMA2 Related Muscular Dystrophy (Laminin Alpha 2 related dystrophy/MDC1A/Merosin deficient) LMNA Related Muscular Dystrophy (Laminopathy/LaminA/C, L-CMD, Emery Dreifuss muscular dystrophy) RYR1 Related Myopathy (with dystrophic presentation, including Malignant Hyperthermia, Exertional Myalgia with or without Rhabdomyolysis) SEPN1 Related Myopathy (Rigid Spine Muscular Dystrophy/RSMD1, Congenital Fiber Type Disproportion, Mallory Weiss Body Desmin, Multi-minicore Myopathy) SYNE1 (Nesprin Related Muscular Dystrophy) Telethonin Related Muscular Dystrophy (TCAP/Titin-Cap) Congenital Muscular Dystrophy Not Otherwise Specified (including Merosin Positive) Titin Related LGMD/CMD, LGMD2J Actin Aggregation Myopathy Cap Disease Central Core Disease (including Malignant Hyperthermia, Exertional Myalgia with or without Rhabdomyolysis) Centronuclear Myopathy (including Malignant Hyperthermia, Exertional Myalgia with or without Rhabdomyolysis) Congenital Fiber Type Disproportion (including Malignant Hyperthermia, Exertional Myalgia with or without Rhabdomyolysis) Core Rod Myopathy Hyaline Body Myopathy Multiminicore Myopathy Myotubular Myopathy Nemaline Myopathy Reducing Body Myopathy RYR1 Related Myopathy (including Malignant Hyperthermia, Exertional Myalgia with or without Rhabdomyolysis) Spheroid Body Myopathy Titin Related Myopathy, Titin Related Dialated Cardiomyopathy, LGMD2J Tubular Aggregate Myopathy Zebra Body Disease Myopathy Congenital Myopathy Not Otherwise Specified Congenital Myasthenic Syndrome Escobar Syndrome Myofibrillar Myopathy

Exclusion Criteria:

Charcot Marie Tooth Duchenne/Becker Muscular Dystrophy Facioscapulohumeral Dystrophy/FSHD Kennedy's Disease LGMD-1A (TTID) LGMD-1C (CAV3, Caveloin 3, Caveolinopathy, LQT9, VIP21) LGMD-1D (7q) LGMD-1E (6q23) LGMD-1F (7q32.1-q32.2) LGMD-1G (4q21) LGMD-2A (CAPN3/Calpainopathy) LGMD-2B (DYSF/Dysferlinopathy/Miyoshi Myopathy) LGMD-2C (SGCG) LGMD-2D (SGCA) LGMD-2E (SGCB) LGMD-2F (SGCD) LGMD-2L (AN05/Anoctamin 5) Lipodystrophy Myotonic Dystrophy Oculopharyngeal Muscular Dystrophy Spinal Muscular Atrophy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants in CMDPROS will be selected from the CMD International Registry (CMDIR) based on the inclusion criteria above.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2009-09 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Congenital Muscle Disease Patient and Proxy Reported Outcomes | 10 years
  Correlation between genetic and biopsy findings and their relation to phenotypic and adverse event data.

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Dziewczapolski, PhD, Study Chair — CureCMD, CMDIR
Locations (1):
- Congenital Muscle Disease International Registry (www.cmdir.org), Lakewood, California, United States

REFERENCES:
- [Background] Bonnemann CG, Rutkowski A, Mercuri E, Muntoni F; CMD Outcomes Consortium. 173rd ENMC International Workshop: congenital muscular dystrophy outcome measures 5-7 March 2010, Naarden, The Netherlands. Neuromuscul Disord. 2011 Jul;21(7):513-22. doi: 10.1016/j.nmd.2011.04.004. Epub 2011 Jun 8. No abstract available. PMID 21641800
- [Background] Wang CH, Bonnemann CG, Rutkowski A, Sejersen T, Bellini J, Battista V, Florence JM, Schara U, Schuler PM, Wahbi K, Aloysius A, Bash RO, Beroud C, Bertini E, Bushby K, Cohn RD, Connolly AM, Deconinck N, Desguerre I, Eagle M, Estournet-Mathiaud B, Ferreiro A, Fujak A, Goemans N, Iannaccone ST, Jouinot P, Main M, Melacini P, Mueller-Felber W, Muntoni F, Nelson LL, Rahbek J, Quijano-Roy S, Sewry C, Storhaug K, Simonds A, Tseng B, Vajsar J, Vianello A, Zeller R; International Standard of Care Committee for Congenital Muscular Dystrophy. Consensus statement on standard of care for congenital muscular dystrophies. J Child Neurol. 2010 Dec;25(12):1559-81. doi: 10.1177/0883073810381924. Epub 2010 Nov 15. PMID 21078917
- [Background] Sparks SE, Quijano-Roy S, Harper A, Rutkowski A, Gordon E, Hoffman EP, Pegoraro E. Congenital Muscular Dystrophy Overview - RETIRED CHAPTER, FOR HISTORICAL REFERENCE ONLY. 2001 Jan 22 [updated 2012 Aug 23]. In: Adam MP, Bick S, Mirzaa GM, Pagon RA, Wallace SE, Amemiya A, editors. GeneReviews(R) [Internet]. Seattle (WA): University of Washington, Seattle; 1993-2026. Available from http://www.ncbi.nlm.nih.gov/books/NBK1291/ PMID 20301468
- [Background] Geranmayeh F, Clement E, Feng LH, Sewry C, Pagan J, Mein R, Abbs S, Brueton L, Childs AM, Jungbluth H, De Goede CG, Lynch B, Lin JP, Chow G, Sousa Cd, O'Mahony O, Majumdar A, Straub V, Bushby K, Muntoni F. Genotype-phenotype correlation in a large population of muscular dystrophy patients with LAMA2 mutations. Neuromuscul Disord. 2010 Apr;20(4):241-50. doi: 10.1016/j.nmd.2010.02.001. Epub 2010 Mar 6. PMID 20207543
- [Background] Sewry CA, Jimenez-Mallebrera C, Muntoni F. Congenital myopathies. Curr Opin Neurol. 2008 Oct;21(5):569-75. doi: 10.1097/WCO.0b013e32830f93c7. PMID 18769251
- [Background] Klein A, Clement E, Mercuri E, Muntoni F. Differential diagnosis of congenital muscular dystrophies. Eur J Paediatr Neurol. 2008 Sep;12(5):371-7. doi: 10.1016/j.ejpn.2007.10.002. Epub 2007 Dec 3. PMID 18588847
- [Background] Godfrey C, Clement E, Mein R, Brockington M, Smith J, Talim B, Straub V, Robb S, Quinlivan R, Feng L, Jimenez-Mallebrera C, Mercuri E, Manzur AY, Kinali M, Torelli S, Brown SC, Sewry CA, Bushby K, Topaloglu H, North K, Abbs S, Muntoni F. Refining genotype phenotype correlations in muscular dystrophies with defective glycosylation of dystroglycan. Brain. 2007 Oct;130(Pt 10):2725-35. doi: 10.1093/brain/awm212. Epub 2007 Sep 18. PMID 17878207
- [Background] Ramelli GP, Aloysius A, King C, Davis T, Muntoni F. Gastrostomy placement in paediatric patients with neuromuscular disorders: indications and outcome. Dev Med Child Neurol. 2007 May;49(5):367-71. doi: 10.1111/j.1469-8749.2007.00367.x. PMID 17489811
- [Background] Mellies U, Dohna-Schwake C, Voit T. Respiratory function assessment and intervention in neuromuscular disorders. Curr Opin Neurol. 2005 Oct;18(5):543-7. doi: 10.1097/01.wco.0000180662.03544.5f. PMID 16155437
- [Background] Takaso M, Nakazawa T, Imura T, Okada T, Ueno M, Saito W, Takahashi K, Yamazaki M, Ohtori S. Surgical correction of spinal deformity in patients with congenital muscular dystrophy. J Orthop Sci. 2010 Jul;15(4):493-501. doi: 10.1007/s00776-010-1486-9. Epub 2010 Aug 19. PMID 20721717
- [Background] Schara U, Kress W, Bonnemann CG, Breitbach-Faller N, Korenke CG, Schreiber G, Stoetter M, Ferreiro A, von der Hagen M. The phenotype and long-term follow-up in 11 patients with juvenile selenoprotein N1-related myopathy. Eur J Paediatr Neurol. 2008 May;12(3):224-30. doi: 10.1016/j.ejpn.2007.08.011. Epub 2007 Oct 22. PMID 17951086
- [Background] Nadeau A, Kinali M, Main M, Jimenez-Mallebrera C, Aloysius A, Clement E, North B, Manzur AY, Robb SA, Mercuri E, Muntoni F. Natural history of Ullrich congenital muscular dystrophy. Neurology. 2009 Jul 7;73(1):25-31. doi: 10.1212/WNL.0b013e3181aae851. PMID 19564581
- [Background] van den Engel-Hoek L, Erasmus CE, de Swart BJ, Sie LT, de Groot IJ. Neonatal swallowing assessment and practical recommendations for oral feeding in a girl with a severe congenital myopathy. J Child Neurol. 2011 Aug;26(8):1041-4. doi: 10.1177/0883073811402071. Epub 2011 May 3. PMID 21540369
- [Background] Saito Y, Komaki H, Hattori A, Takeuchi F, Sasaki M, Kawabata K, Mitsuhashi S, Tominaga K, Hayashi YK, Nowak KJ, Laing NG, Nonaka I, Nishino I. Extramuscular manifestations in children with severe congenital myopathy due to ACTA1 gene mutations. Neuromuscul Disord. 2011 Jul;21(7):489-93. doi: 10.1016/j.nmd.2011.03.004. Epub 2011 Apr 21. PMID 21514153
- See also: Related Info — http://www.cmdir.org